CLINICAL TRIAL: NCT06462937
Title: The SPARK Trial: a Digital Exercise Intervention in Patients With Spondyloarthritis
Brief Title: A Digital Exercise Intervention in Patients With Spondyloarthritis
Acronym: SPARK
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Diakonhjemmet Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: DS00735
Record Dates: First submitted 2024-05-13; First posted 2024-06-17 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Spondyloarthritis; Exercise
Keywords: Remote; Digital; High intensity interval training
MeSH Terms: conditions — Spondylarthritis; Motor Activity | interventions — Exercise; Organization and Administration

STUDY DESIGN:
Intervention Model Description: Baseline: randomization to intervention (Exercise) or control (Usual care) 1:1.
  3 months: randomization to intervention (Exercise remotely delivered plan with personalised weekly follow-up) or control (Exercise remotely delivered plan without weekly follow-up)
Who Masked: Care Provider, Outcomes Assessor
Masking Description: The randomization is performed by a study personnel not involved in data collection. Patients are asked not to inform their care-giver or the physiotherapist who perform the study tests which group the patient is allocated to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Exercise with personal supervision 0-3 months (Experimental): Exercise
  Interventions: Behavioral: Exercise with supervision
- Control 0-3 months (No Intervention): Usual care
- Exercise with personal supervision 3-6 months (Experimental): Exercise
  Interventions: Behavioral: Exercise with supervision
- Exercise without personal supervision 3-6 months (Active Comparator): Exercise
  Interventions: Behavioral: Exercise without supervision

INTERVENTIONS:
Behavioral: Exercise with supervision — Remote exercise will be administered with digital supervision. The Exercise group will receive a personalised program with individual adaptations aiming to perform 3 exercise sessions per week including HIIT, strength exercise and moderate intensive aerobic exercise. Participants will consult their rheumatologist parallel to the SPARK trial.
  Arms: Exercise with personal supervision 0-3 months; Exercise with personal supervision 3-6 months
Behavioral: Exercise without supervision — Remote exercise will be administered without digital supervision. Participants will receive a standard exercise program fulfilling the exercise protocol requirements, the exercise program will progress. But there will be no direct contact between the participant and the coach. Participants will consult their rheumatologist parallel to the SPARK trial.
  Arms: Exercise without personal supervision 3-6 months

SUMMARY:
This protocol describes a 6-month randomised, controlled exercise trial in patients with axial spondyloarthritis (axSpA) with re-randomization after 3-months. The primary outcome of the trial (disease activity) will be evaluated at 3-months. The exercise programme on trial comprises high intensity interval training (HIIT), muscular strength exercise and aerobic physical activity sessions of specified duration, frequency, and intensity. It also includes brief knowledge videos to empower the patient. The intervention is remotely delivered by the SPARK application with personalised follow-up including monitoring to ensure exercise progression and adherence to exercise intensity. The SPARK application is built on a platform delivered by ABEL Technologies (trademark) and is customised for patients with axSpA.

DETAILED DESCRIPTION:
Main objectives: To assess if a digital personally tailored exercise program with remote follow-up can reduce disease activity measured by ankylosing spondylitis disease activity score (ASDAS) in patients with recently diagnosed axial spondyloarthritis (axSpA).

Main inclusion criteria Adults (> 18 years) with clinical diagnosis from a rheumatologist of axSpA within the last 2 years of inclusion also fulfilling the ankylosing spondylitis disease activity score (ASAS) classification criteria, who are biologic disease modifying anti-rheumatic drugs (bDMARD) naïve, and have an active disease (ASDAS ≥ 1.3)

Main exclusion criteria:

Active iridocyclitis, c-reactive protein (CRP) > 30, contraindication to high intensity interval training

Primary outcome Proportion of participants in ASDAS inactive (ASDAS < 1.3) at 3 months

Number of participants: 260 (with an anticipated drop-out rate of 15%)

Study design: A two-arm multi-centre, clinical trial, randomization 1:1 to either digital exercise intervention with remote follow-up or usual care.

Intervention: Exercise delivered through an application and with personalised follow-up by a coach through remote sessions (the participant and SPARK-coach are not at the same physical location) weekly. The exercise is progressively tailored to the fitness level of each participant. The program consists of 5 session per week on 3 different days including: two sessions with HIIT, 2 sessions with strength exercise, and one session with an aerobic exercise at moderate intensity. Goal for HIIT is 10 minutes two times per week at 85-95% of maximal heart rate (20 minutes in total). The exercise will be performed at a location of the participants' choice and data will be logged by a sports watch.

Efficacy assessments: ASDAS disease activity measure (4 patient reported questions and measure of CRP), Bath ankylosing spondylitis disease activity index (BASDAI).

Physical measure: cardiorespiratory fitness, in a subset of participants direct cardiopulmonary testing, muscular strength tests.

Psychological measures: Warwick and Edinburgh mental wellbeing scale (WEMWBS), EuroQol (EQ5D).

Medication: use of bDMARDs, use of NSAID

Safety assessments General physical examination and vital signs, laboratory tests as a part of usual clinical care, record of adverse events and serious adverse events, magnetic resonance imaging (MRI).

ELIGIBILITY:
Inclusion Criteria:

* axSpA diagnosis within the last two years by a rheumatologist according to the ASAS criteria of 2009
* active disease (ASDAS > 1.3)

Exclusion Criteria:

* Active uveitis.
* CRP > 30.
* Former or current use of bDMARDs.
* Pregnancy or planned pregnancy within 6 months from inclusion.
* Absolute and relative contradictions to high intensity exercise according to the American College of Sports Medicine (ACSM)
* Other serious disease such as cancer.
* Patients incapable to follow the protocol or the control set-up with remote monitoring.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2027-08-01 (Estimated); Study Completion 2030-08-01 (Estimated)

PRIMARY OUTCOMES:
Disease activity 3 months | 3 months
  Number of participants in ASDAS inactive (ASDAS < 1.3) at 3 months

SECONDARY OUTCOMES:
Biologic disease modifying anti-rheumatic drugs 3 months | 3 months
  Number of participants on biologic disease modifying anti-rheumatic drugs (bDMARD) at 3 months
Disease activity 6 months | 6 months
  Number of participants in ankylosing spondylitis disease activity score (ASDAS) inactive (ASDAS < 1.3) at 6 months
Proportion of participants using non-steroidal anti-inflammatory drugs | 3 and 6 months
  Usage of non-steroidal anti-inflammatory drugs (NSAIDs)
Bath ankylosing spondylitis metrology index | 3 and 6 months
  Physical function measured by Bath ankylosing spondylitis metrology index (BASMI). Range 0-10 where 0= no functional impairment 10=very significant impairment
Bath ankylosing spondylitis function index | 3 and 6 months
  Physical function measured by Bath ankylosing spondylitis function index (BASFI). Scale range 0-10, where 0= no functional impairment 10=very significant impairment
Ankylosing spondylitis Performance Index | 3 and 6 months
  Physical function measured by Ankylosing spondylitis Performance Index (ASPI). Continuous variable in units of minutes. The functional level is inversely proportional to the number of minutes.
Physical fitness | 3 and 6 months
  Indirect exercise test on a tread-mill until exhaustion. Measured in oxygen uptake ml/min/kg.
Physiological effects of exercise on lipids | 3 and 6 months
  Effect of exercise on lipids
Physiological effects of exercise on inflammation measured by CRP | 3 and 6 months
  Effect of exercise on CRP
Physiological effects of exercise on blood pressure | 3 and 6 months
  Effect of exercise on blood pressure
Physiological effects of exercise on weight | 3 and 6 months
  Effect of exercise on weight in kg
Physiological effects of exercise on muscle mass | 3 and 6 months
  Effect of exercise on body composition measured as percentage muscle mass
Physiological effects of exercise on adipose tissue | 3 and 6 months
  Effect of exercise on body composition measured as percentage adipose tissue
Safety measures of exercise Spine | 3 and 6 months
  Safety measures: MRI spine in a subset of participants at baseline and after 3 months of exercise. Level of inflammation scored by Canadian Spondyloarthritis Research Consortium score (SPARCC). High score represents more inflammation. The minimum score 0, max score 108
Safety measures of exercise Sacroiliac joints | 3 and 6 months
  Safety measures: MRI sacroiliac joints in a subset of participants at baseline and after 3 months of exercise. Level of inflammation scored by Canadian Spondyloarthritis Research Consortium (SPARCC). High score represents more inflammation. The minimum score 0, max score 72
Effects of exercise on mental wellbeing | 3 and 6 months
  Quality of life Warwick Edinburgh Mental Wellbeing Scale WEMWBS). Range 14-70. A higher score indicates greater mental well-being
Effects of exercise on quality of life | 3 and 6 months
  Quality of life EQ5D. Range -0.59 to 1, where 1 is the best possible health state
Work presenteeism | 3 and 6 months
  Health economy measures: work presenteeism expressed in percentage (%) measured by Work Productivity and Activity Impairment Questionnaire (WPAI)
Work absenteeism | 3 and 6 months
  Health economy measures: work absenteeism expressed in percentage (%) measured by Work Productivity and Activity Impairment Questionnaire (WPAI)
Work impairment | 3 and 6 months
  Health economy measures: work overall impairment expressed in percentage (%) measured by Work Productivity and Activity Impairment Questionnaire (WPAI)
Functional impairment | 3 and 6 months
  Health economy measures: functional impairment expressed in percentage (%) measured by Work Productivity and Activity Impairment Questionnaire (WPAI)
Contact with the Healthcare services | 3 and 6 months
  Health economy measures: Contact with the health care services. Self reported as number of visits to general practitioner, specialist healthcare and/or physiotherapist during past 3 months
Sleep quality | 3 and 6 months
  Questionnaire on sleep quality: Pittsburgh Sleep Questionnaire. Global score ranges from 0 to 21 and higher scores indicate poorer sleep quality.
Physical activity level | Baseline, 3 and 6 months
  Physical activity level measured for one week at baseline, 3 months and 6 months by a movement sensor. (Actigraph). The score will be presented as Metabolic Equivalents. A high score represents more movement

CONTACTS AND LOCATIONS:
Locations (1):
- Diakonhjemmet hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No